CLINICAL TRIAL: NCT02171039
Title: Relative Bioavailability of Dabigatran and Atorvastatin After 150 mg BID Dabigatran Etexilate and Atorvastatin at 80 mg QD Alone or Following Concomitant Multiple Oral Administrations in Healthy Male and Female Volunteers (an Open-label, Randomised, Multiple-dose, Three-way Crossover Study)
Brief Title: Relative Bioavailability of Dabigatran and Atorvastatin in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.58
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Atorvastatin

ARMS (3):
- dabigatran plus atorvastatin (Experimental)
  Interventions: Drug: Dabigatran; Drug: Atorvastatin
- dabigatran (Active Comparator)
  Interventions: Drug: Dabigatran
- atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Dabigatran
  Arms: dabigatran; dabigatran plus atorvastatin
Drug: Atorvastatin
  Arms: atorvastatin; dabigatran plus atorvastatin

SUMMARY:
To investigate the bioavailability of dabigatran with and without concomitant administration of atorvastatin and the bioavailability of atorvastatin with and without concomitant administration of dabigatran etexilate

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥18 and ≤65 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Liver transaminases (ALT; aspartate aminotransferase (AST); GGT) and creatin kinase (CK) are to be within the normal range
5. Haemoglobin values within the normal range
6. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Relevant surgery of gastrointestinal tract
3. History of any bleeding disorder or acute blood coagulation defect
4. History or presence of acute liver disease
5. History or presence of myopathy
6. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
7. History of relevant orthostatic hypotension, fainting spells or blackouts
8. Chronic or relevant acute infections
9. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
10. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
11. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
12. Participation in another trial with an investigational drug within two months prior to administration or during the trial
13. Alcohol abuse (more than 60 g/day)
14. Drug abuse
15. Within 5 days of study medication no intake of grapefruit, grapefruit juice, or products containing grapefruit juice, Seville oranges, garlic supplements, or St. John's Wort
16. Blood donation (more than 100 mL within four weeks prior to administration o during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of study centre
20. Females of child bearing potential who are pregnant, breast feeding or who are either not surgically sterile or are sexually active and not using an acceptable form of contraception as either the oral contraceptives since at least two months or the double barrier method, i.e. intrauterine device with spermicide and condom for the male partner
21. Male subjects will not agree to minimise the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the post study medical. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two month)
22. Planned surgeries within four weeks following the end-of study examination
23. Intake of medication, which influences the blood clotting, i.e., acetylsalicylic acid, cumarin etc.
24. The subject is not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
25. Vulnerable subjects (e.g. persons kept in detention).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state over one dosing interval ( AUCτ,ss) | Day 4
Maximum concentration of the analyte in plasma at steady state (Cmax,ss) | 2 hours before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after drug administration on day 4

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma from the time point 0 after the last dose at steady state to the last quantifiable analyte plasma concentration within the uniform dosing interval τ (AUC0-tz,ss) | Up to day 7 after administration
Time of last measurable concentration of the analyte in plasma within the dosing interval τ at steady state (tz,ss) | Up to day 7 after administration
Time from last dosing to the maximum concentration of the analyte in plasma at steady state (tmax,ss) | Up to day 7 after administration
Apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration (CL/Fss) | Up to day 7 after administration
Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | 2 hours before and 0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours after drug administration
Time from last dosing to the minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (tmin,ss ) | Up to day 7 after administration
Pre-dose concentration of the analyte in plasma at steady state immediately before administration of the next dose (Cpre,ss) | 2 hours before drug administration on day 1, 2, 3 and 4
Mean residence time of the analyte in the body at steady state after p.o. administration (MRTp.o.,ss) | Up to day 7 after administration
Apparent volume of distribution during the terminal phase λz at steady state following an extravascular administration (Vz/Fss) | Up to day 7 after administration
Amount of analyte that was eliminated in urine at steady state over an uniform dosing interval τ (Aeτ,ss) | Day 4 and 5 after administration
Fraction of parent drug eliminated in urine at steady state over a uniform dosing interval τ (feτ,ss) | Day 4 and 5 after administration
Renal clearance of the analyte at steady state determined over the dosing interval τ (CLR,ss) | Day 4 and 5 after administration
Maximum effect ratio at steady state (ERmax_ss) for activated thrombin time (aPTT) and ecarin clotting time (ECT) | Up to day 7 after administration
Area under the effect curve (baseline corrected) (AUECτ,ss) for aPTT and ECT | Day 4 and 5
Change from baseline in blood pressure and puls rate (BP, PR) | Baseline, day 78
Change from baseline in physical examination | Baseline, day 78
Change from baseline in 12-lead electrocardiogram | Baseline, day 78
Change from baseline in clinical laboratory tests | Baseline, day 78
Number of Participants with Serious and Non-Serious Adverse Events | Up to day 78
Assessment of tolerability by investigator on a four point scale (good, satisfactory, not satisfactory, bad) | Day 78
Ecarin clotting time (ECT) prolongation at trough (ER(pre,ss)) | Up to day 7 after administration
Amount of total active HMG-CoA reductase inhibitors in plasma | Up to day 7 after administration
Activated partial thromboplastin time (aPTT) prolongation at trough (ER(pre,ss)) | Up to day 7 after administration